CLINICAL TRIAL: NCT00080405
Title: Repeat-Dose Pharmacokinetics and Pharmacodynamics of Bortezomib in Patients With Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M34103-058
Record Dates: First submitted 2004-03-30; First posted 2004-04-02 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-03

CONDITIONS: Multiple Myeloma
Keywords: Relapsed; Multiple Myeloma; Pharmacokinetic; Pharmacodynamic
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Bortezomib

INTERVENTIONS:
Drug: Bortezomib

SUMMARY:
The purpose of this study is to characterize the clinical pharmacokinetic and pharmacodynamic profiles of the 2 doses of VELCADE (bortezomib) for Injection. Patients who volunteer to participate in the pharmacogenetic portion of the study, an additional blood sample will be collected before the Cycle 1 Day 1 dose of bortezomib to assess the genotype of drug metabolizing enzymes.

ELIGIBILITY:
Male and female adult patients 18 years or older with a diagnosis of relapsed multiple myeloma requiring therapy will be eligible for this study.

Key inclusion criteria include:

Karnofsky Performance Status (KPS) equal to or greater then 70%, normal liver function tests (aspartate transaminase [AST] or alanine transaminase [ALT] equal to or less then 2 x upper limit of normal [ULN], total bilirubin equal to or less then 1.5 x ULN), hemoglobin equal to or greater then 10 g/dL, platelets equal to greater then 50 x 10 to ninth power/L, and absolute neutrophil count (ANC) equal to or greater then 1000/uL; calculated creatinine clearance equal to or greater then 50 mL/min, and normal serum calcium.

Key exclusion criteria include:

Patients with significant cardiac disease, equal to or greater then Grade 2 neuropathy, active hepatitis, HIV infection, secondary malignancy, POEMS syndrome, plasma cell leukemia, or who are transfusion-dependent or received extensive radiation therapy, systemic chemotherapy, or other antineoplastic therapy within 4 weeks of enrollment will be excluded. Patients taking concurrent medications at entry that may act as inducers or inhibitors of CYP 3A4 are excluded. Patients receiving thalidomide must discontinue that drug at least 2 weeks prior to enrollment. Patients receiving concurrent corticosteroids must have tapered their dose of corticosteroid to to equal to or less then 10 mg/day of prednisone or prednisone equivalent at least 2 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-03; Primary Completion 2005-06 (Actual)